CLINICAL TRIAL: NCT01394276
Title: Rheumatoid Arthritis Patients Treated With Tocilizumab in Real Clinical Practice: Effectiveness and Safety (TRUST Study)
Brief Title: An Observational Study on RoActemra/Actemra (Tocilizumab) in Clinical Practice in Patients With Rheumatoid Arthritis (TRUST)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25728
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Results first posted 2016-06-07 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Tocilizumab: Participants with moderate to severe Rheumatoid arthritis (RA) who had received RoActemra [Tocilizumab (TCZ)] treatment for 6 months prior to initiation of study and are inadequate responders to Disease Modifying Anti-Rheumatic Drugs (DMARDs) and anti-Tumor Necrosis Factors (anti-TNFs) agents were observed. Participants received treatment with TCZ with dose of 8 milligrams per kilogram (mg/kg) body weight, intravenously once every 4 weeks for 12 months according to European Union (EU) approved dosage, and Summary of Product Characteristics (SmPC).

SUMMARY:
This observational study will evaluate the efficacy and safety of RoActemra/Actemra (tocilizumab) in clinical practice in patients with moderate to severe rheumatoid arthritis. Data will be collected from patients for the 12 months following the first infusion of RoActemra/Actemra.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Rheumatoid arthritis diagnosed according to American College of Rheumatology (ACR) criteria
* Initiated on RoActemra/Actemra treatment according to the Summary of Product Characteristics not more than 6 months before opening of study center

Exclusion Criteria:

* Current serious infection
* Hypersensitivity to the active component or any of the excipients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis initiated on treatment with RoActemra/Actemra
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (48):
- Italy (48):
  - Coppito, Abruzzo
  - Pescara, Abruzzo
  - Brindisi, Apulia
  - Casarano (LE), Apulia
  - Foggia, Apulia
  - Martina Franca, Apulia
  - San Cesario di Lecce, Apulia
  - Reggio Calabria, Calabria
  - Avellino, Campania
  - Gragnano, Campania
  - Napoli, Campania
  - Salerno, Campania
  - Telese Terme, Campania
  - Bologna, Emilia-Romagna
  - Ferrara, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Piacenza, Emilia-Romagna
  - Trieste, Friuli Venezia Giulia
  - Albano Laziale, Lazio
  - Rome, Lazio
  - Viterbo, Lazio
  - Arenzano, Liguria
  - Castel Goffredo, Lombardy
  - Gavardo, Lombardy
  - Legnano, Lombardy
  - Milan, Lombardy
  - Monza, Lombardy
  - Pavia, Lombardy
  - Rozzano, Lombardy
  - Saronno, Lombardy
  - Treviglio, Lombardy
  - Vimercate, Lombardy
  - Agnone, Molise
  - Cuneo, Piedmont
  - Novara, Piedmont
  - Turin, Piedmont
  - Sassari, Sardinia
  - Catania, Sicily
  - Gazzi, Sicily
  - Palermo, Sicily
  - Ancona, The Marches
  - Iesi, The Marches
  - Florence, Tuscany
  - Massa, Tuscany
  - Pisa, Tuscany
  - Prato, Tuscany
  - Perugia, Umbria
  - Verona, Veneto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 322 participants were enrolled across 59 study centers in Italy from 31 May 2011 to 24 April 2013.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 322
Completed | 260
Not Completed | 62
Not completed — Related Adverse event (AEs) | 15
Not completed — Not related AEs | 9
Not completed — Remission of disease | 2
Not completed — Insufficient therapeutic effect | 17
Not completed — Insufficient compliance | 9
Not completed — Lost to Follow-up | 5
Not completed — Participant moved to another site | 1
Not completed — Pregnancy | 1
Not completed — unavailability of drug at the Hospital | 2
Not completed — Symptoms of concurrent diseases | 1

BASELINE CHARACTERISTICS:
Population: The total population included all participants who met all inclusion/exclusion criteria described in the study and received at least one dose of study medication.
Groups:
- Tocilizumab: Participants with moderate to severe RA who had received TCZ treatment for 6 months prior to initiation of study and are inadequate responders to DMARDs and anti-TNFs agents were observed. Participants received treatment with TCZ with dose of 8 mg/kg body weight, intravenously once every 4 weeks for 12 months according to EU approved dosage, and SmPC.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 260
  Male | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Low Disease Activity After 6 Months of Treatment
Description: Low disease activity is defined as a disease activity score based on 28 joint count (DAS28) score lesser or equal to (</=) 3.2. The DAS28 is an evaluation index of RA. DAS28 applies a mathematical formula based on the following parameters: 1. Tender joints count (28 joints), 2. Swollen joints count (28 joints), 3. Erythrocyte sedimentation rate (ESR) or C reactive protein (CRP) measurement, 4. Participant's judgement on his own overall health status expressed by a visual analogue scale (VAS). The DAS28 scale ranges from 0 to 10, where scores below 2.6 indicate best disease control, scores above 5.1 indicate worse disease control, higher scores represent higher disease activity and negative change from baseline score indicates improvement. Percentage of participants with low disease activity was reported.
Time Frame: Up to 12 months
Population: The total population included all participants who met all inclusion/exclusion criteria described in the study and received at least one dose of study medication. Data allowing the evaluation of low disease activity was available for 226 participants in TCZ group.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 226
percentage of participants | 57.52
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p = 0.0237, Exact binomial proportion test

2. Primary Outcome: Percentage of Participants Achieving Disease Remission After 6 Months of Treatment
Description: Disease remission is defined as a DAS28 score < 2.6. The DAS28 is an evaluation index of RA. DAS28 applies a mathematical formula based on the following parameters: 1. Tender joints count (28 joints), 2. Swollen joints count (28 joints), 3. ESR or CRP measurement, 4. Participant's judgment on his own overall health status expressed by a VAS and calculates total score of 0 to approximately 10. The DAS28 scale ranges from 0 to 10, where scores below 2.6 indicate best disease control, scores above 5.1 indicate worse disease control, higher scores represent higher disease activity and negative change from baseline score indicates improvement. The response to therapy is defined according to the disease activity detected, compared to the previous clinical evaluation. Percentage of participants with disease remission was reported.
Time Frame: Up to 12 months
Population: The total population included all participants who met all inclusion/exclusion criteria described in the study and received at least one dose of study medication. Data allowing the evaluation of disease remission was available for 226 participants in TCZ group.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 226
percentage of participants | 38.05
Statistical Analysis 1: Comparison: Tocilizumab; Test type: Superiority or Other; p = 0.0003, Exact binomial proportion test

3. Secondary Outcome: Mean Score of Disease Activity Based on 28 Joint Count in Participants on Monotherapy With Tocilizumab
Description: The DAS28 is an evaluation index of RA. DAS28 applies a mathematical formula based on the following parameters: 1. Tender joints count (28 joints), 2. Swollen joints count (28 joints), 3.ESR or CRP measurement, 4. Participant's judgment on his own overall health status expressed by a VAS and calculates total score of 0 to approximately 10. The DAS28 scale ranges from 0 to 10, where scores below 2.6 indicate best disease control, scores above 5.1 indicate worse disease control, higher scores represent higher disease activity and negative change from baseline score indicates improvement. The response to therapy is defined according to the disease activity detected, compared to the previous clinical evaluation.
Time Frame: Baseline (Month 0), Month 1, Month 2, Month 4, Month 6, and Month 12
Population: The total population included all participants who met all inclusion/exclusion criteria described in the study and received at least one dose of study medication. Data allowing the evaluation of disease activity based on 28 joints count was available for 93 participants in TCZ group. The "n" represents the number of participants analyzed at a specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 93
units on a scale
  Baseline; n = 93 | 5.4 (1.3)
  Month 1; n = 60: number analyzed (Participants) | 60
  Month 1; n = 60 | 3.6 (1.3)
  Month 2; n = 63: number analyzed (Participants) | 63
  Month 2; n = 63 | 3.3 (1.1)
  Month 4; n = 64: number analyzed (Participants) | 64
  Month 4; n = 64 | 3.2 (1.3)
  Month 6; n = 75: number analyzed (Participants) | 75
  Month 6; n = 75 | 3.0 (1.2)
  Month 12; n = 61: number analyzed (Participants) | 61
  Month 12; n = 61 | 2.8 (1.2)

4. Secondary Outcome: Mean Score of Fatigue Based on Visual Analogue Scale in Participants on Monotherapy With Tocilizumab
Description: VAS for fatigue is a 100 mm scale for participant's assessment of their current level of fatigue. The '0 'mm corresponds to "no perception of fatigue," '100 mm' is the "maximum level of fatigue that may be perceived." Mean score of VAS fatigue in participants were reported.
Time Frame: Baseline, Month 1, Month 2, Month 4, Month 6, and Month 12
Population: The total population included all participants who met all inclusion/exclusion criteria described in the study and received at least one dose of study medication. Data allowing the evaluation of fatigue based on VAS was available for 50 participants in TCZ group. The "n" represents the number of participants analyzed at a specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 50
units on a scale
  Baseline; n = 50 | 62.8 (23.2)
  Month 1; n = 39: number analyzed (Participants) | 39
  Month 1; n = 39 | 48.2 (27.9)
  Month 2; n = 36: number analyzed (Participants) | 36
  Month 2; n = 36 | 41.8 (25.6)
  Month 4; n = 39: number analyzed (Participants) | 39
  Month 4; n = 39 | 38.8 (26.6)
  Month 6; n = 48: number analyzed (Participants) | 48
  Month 6; n = 48 | 38.8 (26.1)
  Month 12; n = 46: number analyzed (Participants) | 46
  Month 12; n = 46 | 33.1 (24.9)

5. Secondary Outcome: Mean Score of Health Assessment Questionnaire in Participants on Monotherapy With Tocilizumab
Description: The health assessment questionnaire (HAQ) is a participant-completed questionnaire specific for RA, recommended by the American college of Rheumatology for the evaluation of quality of life. It consists of 20 questions referring to 8 component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities. There are 4 possible responses for each question: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, 3 = unable to do. To calculate HAQ, the participant must have a component set score for at least 6 of 8 component set. The HAQ is the sum of the scores, divided by the number of component set that have a score (in range 6-8) for a total possible score of minimum/maximum i.e., 0 (best) to 3 (worst).
Time Frame: Baseline, Month 1, Month 2, Month 4, Month 6, and Month 12
Population: The total population included all participants who met all inclusion/exclusion criteria described in the study and received at least one dose of study medication. Data allowing the evaluation of HAQ was available for 66 participants in TCZ group. The "n" represents the number of participants analyzed at a specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 66
units on a scale
  Baseline; n = 66 | 1.6 (0.8)
  Month 1; n = 50: number analyzed (Participants) | 50
  Month 1; n = 50 | 1.2 (0.7)
  Month 2; n = 55: number analyzed (Participants) | 55
  Month 2; n = 55 | 1.1 (0.8)
  Month 4; n = 54: number analyzed (Participants) | 54
  Month 4; n = 54 | 1.0 (0.9)
  Month 6; n = 59: number analyzed (Participants) | 59
  Month 6; n = 59 | 1.1 (0.8)
  Month 12; n = 50: number analyzed (Participants) | 50
  Month 12; n = 50 | 1.1 (0.8)

6. Secondary Outcome: Number of Participants With Concomitant Medications
Description: Number of participants treated with at least one concomitant medication i.e., corticosteroid (Prednisone, Methyl prednisolone) was reported.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 322
participants
  Prednisone | 142
  Methylprednisolone | 130

7. Secondary Outcome: Percentage of Participants Discontinuing Treatment With Tocilizumab
Description: The percentage of participants who prematurely discontinued treatment with TCZ during the study period was reported.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 322
percentage of participants | 19.2

8. Secondary Outcome: Number of Participants With Any Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. A Serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 322
participants
  Any AE | 214
  Any SAE | 28

9. Secondary Outcome: Percentage of Participants Still on Tocilizumab Treatment Till 12 Months After the 1st Infusion
Description: Percentage of participants who continued treatment till 12 months after the first infusion with TCZ was reported.
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 322
percentage of participants | 80.8

10. Secondary Outcome: Number of Participants With Presence and Severity of Synovial Hyperplasia, Joint Effusion and Vascularisation of Second Metacarpo-phalangeal Joint of Right Hand.
Description: The presence and severity of synovial hyperplasia (SH) and joint effusion (JE) of second metacarpo-phalangeal (MCP) joint of right hand was determined by ultrasound examination. According to the method proposed by Naredo, synovial hyperplasia and joint effusion were evaluated based on scoring from 1 to 3 (1 = mild, 2 = moderate, 3 = marked). Vascularization was evaluated with power doppler ultrasound and the score was assessed by a semi quantitative scale ranging from 0 to 3 (0 = normal; 1 = slight, evidence of a single flow signal; 2 = moderate, confluent vessels; 3 = marked, evidence of multiple flow signals in over half the intra articular surface).
Time Frame: Baseline, Month 1, Month 2, Month 4, Month 6, and Month 12
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 322
participants
  SH Absent, Baseline | 25
  SH Mild, Baseline | 7
  SH Moderate, Baseline | 16
  SH Marked, Baseline | 5
  SH Absent, Month 1 | 1
  SH Mild, Month 1 | 1
  SH Moderate, Month 1 | 3
  SH Marked, Month 1 | 1
  SH Absent, Month 2 | 2
  SH, Mild, Month 2 | 3
  SH Moderate, Month 2 | 6
  SH Marked, Month 2 | 0
  SH Absent, Month 4 | 2
  SH Mild, Month 4 | 4
  SH Moderate, Month 4 | 3
  SH Marked, Month 4 | 0
  SH Absent, Month 6 | 4
  SH Mild, Month 6 | 5
  SH Moderate, Month 6 | 4
  SH Marked, Month 6 | 0
  SH Absent, Month 12 | 4
  SH Mild, Month 12 | 6
  SH Moderate, Month 12 | 3
  SH Marked, Month 12 | 0
  JE Absent, Baseline | 23
  JE Mild, Baseline | 9
  JE Moderate, Baseline | 17
  JE Marked, Baseline | 6
  JE Absent, Month 1 | 1
  JE Mild, Month 1 | 1
  JE Moderate, Month 1 | 3
  JE Marked, Month 1 | 1
  JE Absent, Month 2 | 4
  JE Mild, Month 2 | 6
  JE Moderate, Month 2 | 1
  JE Marked, Month 2 | 0
  JE Absent, Month 4 | 3
  JE Mild, Month 4 | 5
  JE Moderate, Month 4 | 2
  JE Marked, Month 4 | 0
  JE Absent, Month 6 | 7
  JE Mild, Month 6 | 5
  JE Moderate, Month 6 | 1
  JE Marked, Month 6 | 0
  JE Absent, Month 12 | 7
  JE Mild, Month 12 | 6
  JE Moderate, Month 12 | 0
  JE Marked, Month 12 | 0
  Vascularization, Absent, Baseline | 26
  Vascularization, Mild, Baseline | 8
  Vascularization, Moderate, Baseline | 8
  Vascularization, Marked, Baseline | 11
  Vascularization, Absent, Month 1 | 2
  Vascularization, Mild, Month 1 | 1
  Vascularization, Moderate, Month 1 | 2
  Vascularization, Marked, Month 1 | 1
  Vascularization, Absent, Month 2 | 4
  Vascularization, Mild, Month 2 | 7
  Vascularization, Moderate, Month 2 | 0
  Vascularization, Marked, Month 2 | 0
  Vascularization, Absent, Month 4 | 2
  Vascularization, Mild, Month 4 | 4
  Vascularization, Moderate, Month 4 | 2
  Vascularization, Marked, Month 4 | 0
  Vascularization, Absent, Month 6 | 6
  Vascularization, Mild, Month 6 | 3
  Vascularization, Moderate, Month 6 | 2
  Vascularization, Marked, Month 6 | 0
  Vascularization, Absent, Month 12 | 12
  Vascularization, Mild, Month 12 | 1
  Vascularization, Moderate, Month 12 | 0
  Vascularization, Marked, Month 12 | 0

11. Secondary Outcome: Number of Participants With Presence and Severity of Synovial Hyperplasia, Joint Effusion and Vascularisation of Third Metacarpo-phalangeal Joint of Right Hand.
Description: The presence and severity of SH and JE of third MCP joint of right hand was determined by ultrasound examination. According to the method proposed by Naredo, SH and JE were evaluated based on scoring from 1 to 3 (1 = mild, 2 = moderate, 3 = marked). Vascularization of third MCP joint of right hand was evaluated with power doppler ultrasound and the score was assessed by a semi quantitative scale ranging from 0 to 3 (0 = normal; 1 = slight, evidence of a single flow signal; 2 = moderate, confluent vessels; 3 = marked, evidence of multiple flow signals in over half the intraarticular surface).
Time Frame: Baseline, Month 1, Month 2, Month 4, Month 6, and Month 12
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 322
participants
  SH Absent, Baseline | 26
  SH Mild, Baseline | 9
  SH Moderate, Baseline | 12
  SH Marked, Baseline | 6
  SH Absent, Month 1 | 2
  SH Mild, Month 1 | 1
  SH Moderate, Month 1 | 2
  SH Marked, Month 1 | 1
  SH Absent, Month 2 | 4
  SH Mild, Month 2 | 7
  SH Moderate, Month 2 | 0
  SH Marked, Month 2 | 0
  SH Absent, Month 4 | 2
  SH Mild, Month 4 | 4
  SH Moderate, Month 4 | 2
  SH Marked, Month 4 | 0
  SH Absent, Month 6 | 6
  SH Mild, Month 6 | 3
  SH Moderate, Month 6 | 2
  SH Marked, Month 6 | 0
  SH Absent, Month 12 | 12
  SH Mild, Month 12 | 1
  SH Moderate, Month 12 | 0
  SH Marked, Month 12 | 0
  JE Absent, Baseline | 26
  JE Mild, Baseline | 7
  JE Moderate, Baseline | 17
  JE Marked, Baseline | 4
  JE Absent, Month 1 | 1
  JE Mild, Month 1 | 1
  JE Moderate, Month 1 | 3
  JE Marked, Month 1 | 1
  JE Absent, Month 2 | 6
  JE Mild, Month 2 | 3
  JE Moderate, Month 2 | 2
  JE Marked, Month 2 | 0
  JE Absent, Month 4 | 4
  JE Mild, Month 4 | 6
  JE Moderate, Month 4 | 0
  JE Marked, Month 4 | 0
  JE Absent, Month 6 | 8
  JE Mild, Month 6 | 4
  JE Moderate, Month 6 | 1
  JE Marked, Month 6 | 0
  JE Absent, Month 12 | 9
  JE Mild, Month 12 | 4
  JE Moderate, Month 12 | 0
  JE Marked, Month 12 | 0
  Vascularization, Absent, Baseline | 27
  Vascularization, Mild, Baseline | 7
  Vascularization, Moderate, Baseline | 8
  Vascularization, Marked, Baseline | 10
  Vascularization, Absent, Month 1 | 2
  Vascularization, Mild, Month 1 | 1
  Vascularization, Moderate, Month 1 | 2
  Vascularization, Marked, Month 1 | 1
  Vascularization, Absent, Month 2 | 4
  Vascularization, Mild, Month 2 | 5
  Vascularization, Moderate, Month 2 | 2
  Vascularization, Marked, Month 2 | 0
  Vascularization, Absent, Month 4 | 4
  Vascularization, Mild, Month 4 | 5
  Vascularization, Moderate, Month 4 | 0
  Vascularization, Marked, Month 4 | 0
  Vascularization, Absent, Month 6 | 8
  Vascularization, Mild, Month 6 | 2
  Vascularization, Moderate, Month 6 | 1
  Vascularization, Marked, Month 6 | 0
  Vascularization, Absent, Month 12 | 12
  Vascularization, Mild, Month 12 | 1
  Vascularization, Moderate, Month 12 | 0
  Vascularization, Marked, Month 12 | 0

12. Secondary Outcome: Number of Participants With Presence and Severity of Synovial Hyperplasia, Joint Effusion and Vascularisation of Second Metacarpo-phalangeal Joint of Left Hand
Description: The presence and severity of SH and JE of second MCP joint of left hand was determined by ultrasound examination. According to the method proposed by Naredo, SH and JE were evaluated based on scoring from 1 to 3 (1 = mild, 2 = moderate, 3 = marked). Vascularization of second MCP joint of left hand was evaluated with power doppler ultrasound and the score was assessed by a semi quantitative scale ranging from 0 to 3 (0 = normal; 1 = slight, evidence of a single flow signal; 2 = moderate, confluent vessels; 3 = marked, evidence of multiple flow signals in over half the intra-articular surface).
Time Frame: Baseline, Month 1, Month 2, Month 4, Month 6, and Month 12
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- Tocilizumab: Participants with moderate to severe RA who had received TCZ treatment for 6 months prior to initiation of study and are inadequate responders to DMARDs and anti-TNFs agents. Participants receiving treatment with TCZ with dose of 8 milligrams mg/kg body weight, intravenously once every 4 weeks for 12 months were observed. Dosage of TCZ was prescribed according to EU approved dosage, and SmPC.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 322
participants
  SH Absent, Baseline | 24
  SH Mild, Baseline | 9
  SH Moderate, Baseline | 16
  SH Marked, Baseline | 3
  SH Absent, Month 1 | 1
  SH Mild, Month 1 | 1
  SH Moderate, Month 1 | 3
  SH Marked, Month 1 | 1
  SH Absent, Month 2 | 2
  SH Mild, Month 2 | 7
  SH Moderate, Month 2 | 2
  SH Marked, Month 2 | 0
  SH Absent, Month 4 | 1
  SH Mild, Month 4 | 5
  SH Moderate, Month 4 | 3
  SH Marked, Month 4 | 0
  SH Absent, Month 6 | 6
  SH Mild, Month 6 | 3
  SH Moderate, Month 6 | 4
  SH Marked, Month 6 | 0
  SH Absent, Month 12 | 6
  SH Mild, Month 12 | 5
  SH Moderate, Month 12 | 2
  SH Marked, Month 12 | 0
  JE Absent, Baseline | 22
  JE Mild, Baseline | 13
  JE Moderate, Baseline | 15
  JE Marked, Baseline | 3
  JE Absent, Month 1 | 1
  JE Mild, Month 1 | 1
  JE Moderate, Month 1 | 3
  JE Marked, Month 1 | 1
  JE Absent, Month 2 | 5
  JE Mild, Month 2 | 5
  JE Moderate, Month 2 | 1
  JE Marked, Month 2 | 0
  JE Absent, Month 4 | 2
  JE Mild, Month 4 | 6
  JE Moderate, Month 4 | 1
  JE Marked, Month 4 | 0
  JE Absent, Month 6 | 8
  JE Mild, Month 6 | 4
  JE Moderate, Month 6 | 1
  JE Marked, Month 6 | 0
  JE Absent, Month 12 | 9
  JE Mild, Month 12 | 4
  JE Moderate, Month 12 | 0
  JE Marked, Month 12 | 0
  Vascularization, Absent, Baseline | 26
  Vascularization, Mild, Baseline | 8
  Vascularization, Moderate, Baseline | 11
  Vascularization, Marked, Baseline | 8
  Vascularization, Absent, Month 1 | 2
  Vascularization, Mild, Month 1 | 1
  Vascularization, Moderate, Month 1 | 2
  Vascularization, Marked, Month 1 | 1
  Vascularization, Absent, Month 2 | 5
  Vascularization, Mild, Month 2 | 6
  Vascularization, Moderate, Month 2 | 0
  Vascularization, Marked, Month 2 | 0
  Vascularization, Absent, Month 4 | 4
  Vascularization, Mild, Month 4 | 3
  Vascularization, Moderate, Month 4 | 2
  Vascularization, Marked, Month 4 | 0
  Vascularization, Absent, Month 6 | 7
  Vascularization, Mild, Month 6 | 3
  Vascularization, Moderate, Month 6 | 1
  Vascularization, Marked, Month 6 | 0
  Vascularization, Absent, Month 12 | 12
  Vascularization, Mild, Month 12 | 1
  Vascularization, Moderate, Month 12 | 0
  Vascularization, Marked, Month 12 | 0

13. Secondary Outcome: Number of Participants With Presence and Severity of Synovial Hyperplasia, Joint Effusion and Vascularisation of Third Metacarpo-phalangeal Joint of Left Hand.
Description: The presence and severity of SH and JE of third MCP joint of left hand was determined by ultrasound examination. According to the method proposed by Naredo, SH and JE were evaluated based on scoring from 1 to 3 (1 = mild, 2 = moderate, 3 = marked). Vascularization of third MCP joint of left hand was evaluated with power doppler ultrasound and the score was assessed by a semi quantitative scale ranging from 0 to 3 (0 = normal; 1 = slight, evidence of a single flow signal; 2 = moderate, confluent vessels; 3 = marked, evidence of multiple flow signals in over half the intra-articular surface).
Time Frame: Baseline, Month 1, Month 2, Month 4, Month 6, and Month 12
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 322
participants
  SH Absent, Baseline | 25
  SH Mild, Baseline | 9
  SH Moderate, Baseline | 14
  SH Marked, Baseline | 5
  SH Absent, Month 1 | 1
  SH Mild, Month 1 | 1
  SH Moderate, Month 1 | 3
  SH Marked, Month 1 | 1
  SH Absent, Month 2 | 2
  SH Mild, Month 2 | 6
  SH Moderate, Month 2 | 3
  SH Marked, Month 2 | 0
  SH Absent, Month 4 | 3
  SH Mild, Month 4 | 4
  SH Moderate, Month 4 | 3
  SH Marked, Month 4 | 0
  SH Absent, Month 6 | 5
  SH Mild, Month 6 | 4
  SH Moderate, Month 6 | 4
  SH Marked, Month 6 | 0
  SH Absent, Month 12 | 8
  SH Mild, Month 12 | 4
  SH Moderate, Month 12 | 1
  SH Marked, Month 12 | 0
  JE Absent, Baseline | 25
  JE Mild, Baseline | 7
  JE Moderate, Baseline | 18
  JE Marked, Baseline | 3
  JE, Absent, Month 1 | 1
  JE Mild, Month 1 | 1
  JE Moderate, Month 1 | 3
  JE Marked, Month 1 | 1
  JE Absent, Month 2 | 5
  JE Mild, Month 2 | 5
  JE Moderate, Month 2 | 1
  JE Marked, Month 2 | 0
  JE Absent, Month 4 | 4
  JE Mild, Month 4 | 6
  JE Moderate, Month 4 | 0
  JE Marked, Month 4 | 0
  JE Absent, Month 6 | 8
  JE Mild, Month 6 | 4
  JE Moderate, Month 6 | 0
  JE Marked, Month 6 | 0
  JE Absent, Month 12 | 11
  JE Mild, Month 12 | 2
  JE Moderate, Month 12 | 0
  JE Marked, Month 12 | 0
  Vascularization, Absent, Baseline | 29
  Vascularization, Mild, Baseline | 8
  Vascularization, Moderate, Baseline | 9
  Vascularization, Marked, Baseline | 7
  Vascularization, Absent, Month 1 | 2
  Vascularization, Mild, Month 1 | 1
  Vascularization, Moderate, Month 1 | 2
  Vascularization, Marked, Month 1 | 1
  Vascularization, Absent, Month 2 | 6
  Vascularization, Mild, Month 2 | 5
  Vascularization, Moderate, Month 2 | 0
  Vascularization, Marked, Month 2 | 0
  Vascularization, Absent, Month 4 | 4
  Vascularization, Mild, Month 4 | 5
  Vascularization, Moderate, Month 4 | 0
  Vascularization, Marked, Month 4 | 0
  Vascularization, Absent, Month 6 | 6
  Vascularization, Mild, Month 6 | 3
  Vascularization, Moderate, Month 6 | 2
  Vascularization, Marked, Month 6 | 0
  Vascularization, Absent, Month 12 | 12
  Vascularization, Mild, Month 12 | 1
  Vascularization, Moderate, Month 12 | 0
  Vascularization, Marked, Month 12 | 0

14. Secondary Outcome: Mean Disease Activity Score Based on 28 Joint Count Score in the Participants With Inadequate Response to Disease Modifying Anti-Rheumatic Drugs and Anti-Tumor Necrosis Factors Agents
Description: The DAS28 index applies a mathematical formula based on the following parameters: 1. Tender joints count (28 joints), 2. Swollen joints count (28 joints) 3. ESR or CRP measurement, 4. Participant's judgment on his own overall health status expressed by a VAS and calculates total score of 0 to approximately 10. The DAS28 scale ranges from 0 to 10, where scores below 2.6 indicate best disease control, scores above 5.1 indicate worse disease control. The response to therapy is defined according to the disease activity detected, compared to the previous clinical evaluation. The mean DAS28 scores were evaluated after the first infusion of TCZ in two different sub populations: participants with inadequate response (IR) to DMARD (DMARD-IR: group A) or to DMARD and anti-TNF drugs (DMARD + anti-TNF-IR: group B). Data allowing the evaluation of DAS28 was available for 81 participants in DMARD-IR group and 203 participants in DMARD + anti-TNF-IR group.
Time Frame: Baseline, Month 1, Month 2, Month 4, Month 6, and Month 12
Population: The total population included all participants who met all inclusion/exclusion criteria described in the study and received at least one dose of study medication. The "n" represents the number of participants analyzed at a specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DMARD-IR: Participants with moderate to severe RA who had received TCZ treatment for 6 months prior to initiation of study and are inadequate responders to DMARDs were observed. Participants received treatment with TCZ with dose of 8 mg/kg body weight, intravenously once every 4 weeks for 12 months according to EU approved dosage, and SmPC.
- DMARD + Anti-TNF-IR: Participants with moderate to severe RA who had received TCZ treatment for 6 months prior to initiation of study and are inadequate responders to DMARDs and anti-TNFs agents were observed. Participants received treatment with TCZ with dose of 8 mg/kg body weight, intravenously once every 4 weeks for 12 months according to EU approved dosage, and SmPC.
Arm/Group | DMARD-IR | DMARD + Anti-TNF-IR
Number analyzed (Participants) | 81 | 203
units on a scale
  Baseline; n = 81, 203 | 5.3 (1.1) | 5.3 (1.3)
  Month 1; n = 54, 150: number analyzed (Participants) | 54 | 150
  Month 1; n = 54, 150 | 3.6 (1.2) | 3.7 (1.3)
  Month 2; n = 62, 144: number analyzed (Participants) | 62 | 144
  Month 2; n = 62, 144 | 3.1 (1.3) | 3.4 (1.3)
  Month 4; n = 64, 127: number analyzed (Participants) | 64 | 127
  Month 4; n = 64, 127 | 3.0 (1.4) | 3.1 (1.2)
  Month 6; n = 65, 158: number analyzed (Participants) | 65 | 158
  Month 6; n = 65, 158 | 3.0 (1.2) | 3.0 (1.2)
  Month 12; n = 60, 125: number analyzed (Participants) | 60 | 125
  Month 12; n = 60, 125 | 2.7 (1.2) | 2.6 (1.1)
Statistical Analysis 1: Comparison: DMARD-IR vs DMARD + Anti-TNF-IR; At Baseline: mean difference of scores of DAS28 between the two groups was calculated; Test type: Superiority or Other; p = 0.8080, t-test, 2 sided; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.3 to 0.4]
Statistical Analysis 2: Comparison: DMARD-IR vs DMARD + Anti-TNF-IR; At Month 1: mean difference of scores of DAS28 between the two groups was calculated; Test type: Superiority or Other; p = 0.4884, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.3]
Statistical Analysis 3: Comparison: DMARD-IR vs DMARD + Anti-TNF-IR; At Month 2: mean difference of scores of DAS28 between the two groups was calculated; Test type: Superiority or Other; p = 0.0947, t-test, 2 sided; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.7 to 0.1]
Statistical Analysis 4: Comparison: DMARD-IR vs DMARD + Anti-TNF-IR; At Month 4: mean difference of scores of DAS28 between the two groups was calculated; Test type: Superiority or Other; p = 0.8181, t-test, 2 sided; Mean Difference (Net) = -0.0, 95% CI 2-sided [-0.4 to 0.3]
Statistical Analysis 5: Comparison: DMARD-IR vs DMARD + Anti-TNF-IR; At Month 6: mean difference of scores of DAS28 between the two groups was calculated; Test type: Superiority or Other; p = 0.9721, t-test, 2 sided; Mean Difference (Net) = -0.0, 95% CI 2-sided [-0.4 to 0.3]
Statistical Analysis 6: Comparison: DMARD-IR vs DMARD + Anti-TNF-IR; At Month 12: mean difference of scores of DAS28 between the two groups was calculated; Test type: Superiority or Other; p = 0.5832, t-test, 2 sided; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.3 to 0.5]

15. Secondary Outcome: Mean Score of Fatigue Based on Visual Analogue Scale in the Participants With Inadequate Response to Disease Modifying Anti-Rheumatic Drugs and Anti-Tumor Necrosis Factors Agents
Description: VAS for fatigue is a 100 mm scale for participant's assessment of their current level of fatigue: 0 mm corresponds to "no perception of fatigue"; 100 mm is the "maximum that may be perceived". The mean VAS fatigue scores were evaluated after the first infusion of TCZ in two different sub populations, classified according to the previous pharmacological treatment: participants with inadequate response to DMARD (DMARD-IR: group A) or to DMARD and anti-TNF drugs (DMARD + anti-TNF-IR: group B). Data allowing the evaluation of fatigue (VAS) was available for 45 participants in DMARD-IR group and 113 participants in DMARD + anti-TNF-IR group.
Time Frame: Baseline, Month 1, Month 2, Month 4, Month 6, and Month 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DMARD- IR: Participants with moderate to severe RA who had received TCZ treatment for 6 months prior to initiation of study and are inadequate responders to DMARDs were observed. Participants received treatment with TCZ with dose of 8 mg/kg body weight, intravenously once every 4 weeks for 12 months according to EU approved dosage, and SmPC.
- DMARD + Anti-TNF- IR: Participants with moderate to severe RA who had received TCZ treatment for 6 months prior to initiation of study and are inadequate responders to DMARDs and anti-TNFs agents were observed. Participants received treatment with TCZ with dose of 8 mg/kg body weight, intravenously once every 4 weeks for 12 months according to EU approved dosage, and SmPC.
Arm/Group | DMARD- IR | DMARD + Anti-TNF- IR
Number analyzed (Participants) | 45 | 113
units on a scale
  Baseline; n = 42, 113: number analyzed (Participants) | 42 | 113
  Baseline; n = 42, 113 | 62.3 (21.6) | 58.7 (25.2)
  Month 1; n = 34, 90: number analyzed (Participants) | 34 | 90
  Month 1; n = 34, 90 | 50.1 (24.2) | 48.0 (25.4)
  Month 2; n = 38, 88: number analyzed (Participants) | 38 | 88
  Month 2; n = 38, 88 | 50.6 (24.0) | 44.1 (25.0)
  Month 4; n = 45, 99: number analyzed (Participants) | 45 | 99
  Month 4; n = 45, 99 | 42.8 (22.9) | 40.0 (24.8)
  Month 6; n = 43, 111: number analyzed (Participants) | 43 | 111
  Month 6; n = 43, 111 | 48.4 (23.6) | 34.7 (25.4)
  Month 12; n = 45, 94: number analyzed (Participants) | 45 | 94
  Month 12; n = 45, 94 | 34.9 (19.9) | 31.0 (24.3)
Statistical Analysis 1: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Baseline: mean difference of scores of fatigue between the two groups was calculated; Test type: Superiority or Other; p = 0.4211, t-test, 2 sided; Mean Difference (Net) = 3.5, 95% CI 2-sided [-5.1 to 12.2]
Statistical Analysis 2: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 1: mean difference of scores of fatigue between the two groups was calculated; Test type: Superiority or Other; p = 0.6749, t-test, 2 sided; Mean Difference (Net) = 2.1, 95% CI 2-sided [-7.9 to 12.1]
Statistical Analysis 3: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 2: mean difference of scores of fatigue between the two groups was calculated; Test type: Superiority or Other; p = 0.1817, t-test, 2 sided; Mean Difference (Net) = 6.4, 95% CI 2-sided [-3.0 to 15.9]
Statistical Analysis 4: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 4: mean difference of scores of fatigue between the two groups was calculated; Test type: Superiority or Other; p = 0.5182, t-test, 2 sided; Mean Difference (Net) = 2.8, 95% CI 2-sided [-5.8 to 11.4]
Statistical Analysis 5: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 6: mean difference of scores of fatigue between the two groups was calculated; Test type: Superiority or Other; p = 0.0025, t-test, 2 sided; Mean Difference (Net) = 13.7, 95% CI 2-sided [4.9 to 22.6]
Statistical Analysis 6: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 12: mean difference of scores of fatigue between the two groups was calculated; Test type: Superiority or Other; p = 0.3540, t-test, 2 sided; Mean Difference (Net) = 3.9, 95% CI 2-sided [-4.4 to 12.1]

16. Secondary Outcome: Mean Score of Health Assessment Questionnaire in the Participants With Inadequate Response to Disease Modifying Anti-Rheumatic Drugs and Anti-Tumor Necrosis Factors Agents
Description: The HAQ is a participant-completed questionnaire specific for RA, recommended by the American college of Rheumatology for the evaluation of quality of life. It consists of 20 questions referring to 8 component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities. There are 4 possible responses for each question: 0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, 3 = unable to do. To calculate HAQ, participant must have a component set score for at least 6 of 8 component set. The HAQ is the sum of the scores, divided by the number of component set that have a score (in range 6-8) for a total possible score minimum/maximum 0 (best) to 3 (worst). Data allowing the evaluation of HAQ was available for 73 participants in DMARD-IR group and 157 participants in DMARD + anti-TNF-IR group.
Time Frame: Baseline, Month 1, Month 2, Month 4, Month 6, and Month 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DMARD- IR | DMARD + Anti-TNF- IR
Number analyzed (Participants) | 73 | 157
units on a scale
  Baseline; n = 73, 157 | 1.5 (0.8) | 1.5 (0.7)
  Month 1; n = 52, 120: number analyzed (Participants) | 52 | 120
  Month 1; n = 52, 120 | 1.1 (0.7) | 1.3 (0.7)
  Month 2; n = 58, 123: number analyzed (Participants) | 58 | 123
  Month 2; n = 58, 123 | 1.2 (0.8) | 1.2 (0.8)
  Month 4; n = 62, 122: number analyzed (Participants) | 62 | 122
  Month 4; n = 62, 122 | 0.9 (0.8) | 1.1 (0.7)
  Month 6; n = 62, 126: number analyzed (Participants) | 62 | 126
  Month 6; n = 62, 126 | 1.0 (0.8) | 1.0 (0.7)
  Month 12; n = 54, 102: number analyzed (Participants) | 54 | 102
  Month 12; n = 54, 102 | 1.0 (0.8) | 0.9 (0.7)
Statistical Analysis 1: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Baseline: mean difference of scores of HAQ between the two groups was calculated; Test type: Superiority or Other; p = 0.7343, t-test, 2 sided; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 2: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 1: mean difference of scores of HAQ between the two groups was calculated; Test type: Superiority or Other; p = 0.1098, t-test, 2 sided; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.0]
Statistical Analysis 3: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 2: mean difference of scores of HAQ between the two groups was calculated; Test type: Superiority or Other; p = 0.4932, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.2]
Statistical Analysis 4: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 4: mean difference of scores of HAQ between the two groups was calculated; Test type: Superiority or Other; p = 0.2468, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.1]
Statistical Analysis 5: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 6: mean difference of scores of HAQ between the two groups was calculated; Test type: Superiority or Other; p = 0.9639, t-test, 2 sided; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 6: Comparison: DMARD- IR vs DMARD + Anti-TNF- IR; At Month 12: mean difference of scores of HAQ between the two groups was calculated; Test type: Superiority or Other; p = 0.6696, t-test, 2 sided; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.3]

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 28/322
Other Adverse Events (participants affected / at risk) | 99/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=322)
Major depression (Psychiatric disorders) | 1
Fibrin D dimer increased (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
Renal abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Hydrocele (Congenital, familial and genetic disorders) | 1
Leucopenia (Blood and lymphatic system disorders) | 1
Hypocomplementaemia (Blood and lymphatic system disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Gynaecomastia (Reproductive system and breast disorders) | 1
Retinal detachment (Eye disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Goitre (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Skin neoplasm excision (Surgical and medical procedures) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=322)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 23
Bronchitis (Infections and infestations) | 23
Influenza (Infections and infestations) | 16
Leucopenia (Blood and lymphatic system disorders) | 20
Neutropenia (Blood and lymphatic system disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.